CLINICAL TRIAL: NCT00073281
Title: Islet Transplantation for Patients With Type 1 Diabetes and Stable Renal Allografts Using Steroid Sparing Immunosuppression
Brief Title: Islet Transplantation for Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9903 (completed)
Record Dates: First submitted 2003-11-18; First posted 2003-11-20 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes; autoimmunity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Autoimmune Diseases | interventions — Islets of Langerhans Transplantation

INTERVENTIONS:
Procedure: Islet transplantation

SUMMARY:
This protocol will test whether Type 1 diabetes (T1DM) can be reversed in patients with stable renal allografts by islet transplantation.

DETAILED DESCRIPTION:
We will test whether pancreatic islets isolated from cadaveric human donor pancreata can be transplanted into the portal vein of patients with T1DM who have stable renal allografts to achieve insulin independence for the recipient. The protocol will employ a defined islet isolation procedure, percutaneous islet infusion into the recipient's portal vein via an intra-portal catheter, tight glycemic control during the peri-transplant period, and an immunosuppressive protocol that avoids glucocorticoids.

ELIGIBILITY:
* Patients with type 1 diabetes with stable renal allografts

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2003-08; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hardy, MD, Principal Investigator — Columbia Presbyterian Hospital
Locations (1):
- Columbia Presbyterian Medical Center, New York, New York, United States